CLINICAL TRIAL: NCT02349282
Title: The Effect of Calcifediol (Hy.D 25 SD/S) and Vitamin D3 on Muscle Strength in a Frail Elderly Population: a Randomized, Double-blind, Placebo-controlled Trial.
Brief Title: The Effect of Calcifediol (Hy.D 25 SD/S) and Vitamin D3 on Muscle Strength in a Frail Elderly Population
Acronym: D-Fit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Top Institute Food and Nutrition (Other); DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL48127.081.148
Record Dates: First submitted 2014-12-22; First posted 2015-01-28 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Deficiency, Vitamin D; Elderly, Frail
Keywords: muscle strength; physical performance; vitamin D3; Cholecalciferol; Calcifediol
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Calcifediol; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Calcifediol 10 ug/day (Experimental): Capsule with 10 ug/day Calcifediol taken together with breakfast for a total period of 24 weeks.
  Interventions: Dietary Supplement: Calcifediol 10ug/day
- Vitamin D3 20 ug/day (Experimental): Capsule with 20 ug/day Vitamin D3 taken together with breakfast for a total period of 24 weeks.
  Interventions: Dietary Supplement: Vitamin D3 20ug/day
- Placebo (Placebo Comparator): Capsule without active ingredients, taken together with breakfast for a total period of 24 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Calcifediol 10ug/day
  Other Names: Hy.D
  Arms: Calcifediol 10 ug/day
Dietary Supplement: Vitamin D3 20ug/day
  Other Names: Cholecalciferol
  Arms: Vitamin D3 20 ug/day
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
In an ageing population, the need for interventions to help older people remain healthy, active and independent for as long as possible, increases. Although several studies suggest a beneficial effect of vitamin D3 on maintaining or improving muscle strength and physical functioning, particularly in vulnerable populations, results are contradicting. Randomized, placebo-controlled trials are needed to further establish the effect of vitamin D on muscle strength in the frail elderly population.The primary aim of this study is to determine the effect of daily supplementation with two different forms of vitamin D on muscle strength in frail elderly people over a period of 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 25(OH)D levels 20-50 nmol/L.
* age 65 or older.
* physically frail (pre-frail or frail, based on the criteria designed by Fried et al.) (30). Frailty will be defined as a clinical syndrome in which one or more of the following criteria are present: unintentional weight loss (4.5 kg in past year), self-reported exhaustion (CES-D questionnaire), weakness (grip strength), slow walking speed and low physical activity (Minnesota questionnaire). More details on these criteria are described in chapter 6.3.2.
* body mass index between 18.5 and 35 kg/m2.
* willingness and ability to comply with the protocol, including performance of the knee extension strength test.

Exclusion Criteria:

* Medical Illness:

  * malabsorption syndrome: known intestinal malabsorption, celiac diseases, inflammatory bowel disease;
  * diseases that may enhance serum calcium concentration: sarcoidosis, lymphoma, kidney stone in the last 10 years, primary hyperparathyroidism;
  * abnormal indices of calcium metabolism, uncontrolled hypocalcaemia;
  * diagnosed renal insufficiency;
  * diagnosed cancer; currently diagnosed or undergoing treatment.
* Hypercalcemia: serum calcium adjusted for albumin of > 2.6 nmol/L.
* Medication: interfering with vitamin D metabolism and vitamin D supplementation (bisphosphonate, PTH treatment, tuberculostatica, anti-epileptica).
* Subject not able (when medically necessary/ advised) or not willing to stop the use of vitamin D containing supplements during the study.
* (Expected) increase in exposure to sunlight (e.g. travelling to a sunny resort) during intervention period.
* Patient heavily consumes alcohol containing products defined as greater than > 21 drinks of alcoholic beverages per week.
* Planned surgery which can affect study measures (taking into account duration of hospitalisation and recovery).
* Participation in another clinical trial.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 78 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in muscle strength, knee extension strength (measured by Biodex System) | baseline, week 12, end of study (after 24 weeks supplementation)
  measured by Biodex System

SECONDARY OUTCOMES:
Change in knee flexion strength (measured by Biodex System) | baseline, week 12, end of study (after 24 weeks supplementation)
  measured by Biodex System
Change in handgrip strength | baseline, week 12, end of study (after 24 weeks supplementation)
Change in SPPB | baseline, week 12, end of study (after 24 weeks supplementation)
Change in Timed Up and Go test | baseline, week 12, end of study (after 24 weeks supplementation)
Change in Postural Body Sway | baseline, week 12, end of study (after 24 weeks supplementation)
Change in serum Vitamin D3 | baseline, week 12, end of study (after 24 weeks supplementation)
Change in serum 25(OH)D | baseline, week 12, end of study (after 24 weeks supplementation)
Change in serum 1,25(OH)2D3 | baseline, week 12, end of study (after 24 weeks supplementation)
Change in serum 24,25(OH)2D | baseline, week 12, end of study (after 24 weeks supplementation)
Frequency of falling | baseline, week 12, end of study (after 24 weeks supplementation)
Change in muscle fibre type and size (Biopsy) | baseline, end of study (after 24 weeks supplementation)
  Biopsy
Change in body composition (DEXA-scan) | baseline, end of study (after 24 weeks supplementation)
  DEXA-scan
Change in cognitive functioning (Trail making, Stroop-test, Letter fluency) | baseline, end of study (after 24 weeks supplementation)
  Trail making, Stroop-test, Letter fluency
Change in vital Signs (blood pressure and heart rate) | baseline, week 12, end of study (after 24 weeks supplementation)
  blood pressure and heart rate
Change in neuromuscular measurements (MUNIX, MUSIX by EMG) | baseline, end of study (after 24 weeks supplementation)
  MUNIX, MUSIX by EMG

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University, Wageningen, Gelderland, Netherlands

REFERENCES:
- [Derived] Hangelbroek RWJ, Vaes AMM, Boekschoten MV, Verdijk LB, Hooiveld GJEJ, van Loon LJC, de Groot LCPGM, Kersten S. No effect of 25-hydroxyvitamin D supplementation on the skeletal muscle transcriptome in vitamin D deficient frail older adults. BMC Geriatr. 2019 May 28;19(1):151. doi: 10.1186/s12877-019-1156-5. PMID 31138136
- [Derived] Vaes AMM, Tieland M, Toussaint N, Nilwik R, Verdijk LB, van Loon LJC, de Groot LCPGM. Cholecalciferol or 25-Hydroxycholecalciferol Supplementation Does Not Affect Muscle Strength and Physical Performance in Prefrail and Frail Older Adults. J Nutr. 2018 May 1;148(5):712-720. doi: 10.1093/jn/nxy024. PMID 30053278